CLINICAL TRIAL: NCT00419471
Title: Efficacy and Safety of Escitalopram in the Treatment of Depressive Patients With Acute Coronary Artery Syndrome: A Double-blind Placebo-controlled Trial
Brief Title: Escitalopram in Depressive Patients With Acute Coronary Artery Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Jae-Min Kim, Associate Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIIS-11592A
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Depressive Disorder; Coronary Disease
Keywords: Depression; Myocardial infarction; Angina, unstable
MeSH Terms: conditions — Depressive Disorder; Coronary Disease; Depression; Myocardial Infarction; Angina, Unstable | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Experimental)
  Interventions: Drug: Escitalopram
- Placebo pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Study medication will be provided as 1 tablet of escitalopram 5mg/day or 1 or 2 tablets of escitalopram 10mg/day, and matched placebo. The initial dose of escitalopram was 10mg/day generally, but 5mg/day for those aged 65 or over and with hepatic dysfunction. After the 2nd evaluation, the treatment doses are determined by the investigators' clinical decision considering the severity of depression and tolerability of drug. Drugs are taken once daily per orally within 30 min after the supper meal.
  Other Names: Lexapro; Cipralex
  Arms: Escitalopram
Drug: Placebo — Placebo medication will be provided as matched 1 tablet of escitalopram 5mg/day or 1 or 2 tablets of escitalopram 10mg/day.
  Arms: Placebo pill

SUMMARY:
This study aimed to evaluate the efficacy and safety of escitalopram in the treatment of depressive patients with acute coronary artery syndrome (CAS).

DETAILED DESCRIPTION:
Depression is common in patients with acute CAS and increases cardiac morbidity and mortality. However, there are a few limited data available regarding the effects and safety of antidepressants for treating depression in patients with acute CAS. This study aims to investigate whether escitalopram might be an effective treatment option for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18~85
* Diagnosed as acute CAS (unstable angina or acute myocardial infarction) and being conducted coronary angiography
* Beck Depression Inventory > 10 and major or minor depressive disorder by the DSM-IV criteria
* With ability to complete various questionnaires
* Can understand the objective of the study and sign informed consent

Exclusion Criteria:

* Occurrence of acute CAS while the patient was hospitalized for another reason, except for CAS
* Current CAS developed less than 3 months after coronary artery bypass graft procedure
* Uncontrolled hypertension (systolic BP > 180mmHg or diastolic BP > 100mmHg)
* Resting heart rate < 40/min
* Severe physical illnesses threatening life or interfering with the recovery from CAS
* Persistent clinically significant laboratory abnormalities
* Concomitant use of class I antiarrhythmic medications; reserpine, guanethidine, clonidine, or methyldopa; anticonvulsants or neuroleptics
* History of neuropsychiatric illnesses such as dementia, Parkinson's disease, brain tumor, psychoses, alcoholism, and other substance dependence
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Score on the Hamilton Depression Rating Scale-17 item | 24 weeks

SECONDARY OUTCOMES:
Scores on the Beck Depression Inventory | 24 weeks
Changes in electrocardiographic, echocardiographic, and angiographic variables | 24 weeks
Scores on the Montgomery Asberg Depression Rating Scale | 24 weeks
Scores on the Clinical Global Impression scale | 24 weeks
Scores on the World Health Organization Quality of Life scale | 24 weeks
Scores on the Social and Occupational Functioning Assessment Scale | 24 weeks
Scores on the World Health Organization Disability Assessment Schedule | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Sang Yoon, MD & PhD, Principal Investigator — Chonnam National University Hospital; Jae-Min Kim, MD & PhD, Study Director — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

REFERENCES:
- [Derived] Choi W, Kim JW, Kang HJ, Kim HK, Kang HC, Lee JY, Kim SW, Hong YJ, Ahn Y, Jeong MH, Stewart R, Kim JM. Interaction effects of diabetes and brain-derived neurotrophic factor on suicidal ideation in patients with acute coronary syndrome. Sci Rep. 2022 Apr 22;12(1):6602. doi: 10.1038/s41598-022-10557-6. PMID 35459929
- [Derived] Kim JW, Stewart R, Lee HJ, Kang HJ, Kim SW, Shin IS, Kim MC, Hong YJ, Ahn YK, Jeong MH, Yoon JS, Kim JM. Sleep problems associated with long-term mortality in acute coronary syndrome: Effects of depression comorbidity and treatment. Gen Hosp Psychiatry. 2020 Sep-Oct;66:125-132. doi: 10.1016/j.genhosppsych.2020.08.004. Epub 2020 Aug 13. PMID 32836109
- [Derived] Kim JM, Stewart R, Kang HJ, Kim SY, Kim JW, Lee HJ, Lee JY, Kim SW, Shin IS, Kim MC, Shin HY, Hong YJ, Ahn Y, Jeong MH, Yoon JS. Long-term cardiac outcomes of depression screening, diagnosis and treatment in patients with acute coronary syndrome: the DEPACS study. Psychol Med. 2021 Apr;51(6):964-974. doi: 10.1017/S003329171900388X. Epub 2020 Jan 7. PMID 31907104
- [Derived] Kim JW, Kang HJ, Bae KY, Kim SW, Shin IS, Yoon JS, Hong YJ, Ahn Y, Jeong MH, Kim JM. Social support deficit and depression treatment outcomes in patients with acute coronary syndrome: Findings from the EsDEPACS study. Int J Psychiatry Med. 2019 Jan;54(1):39-52. doi: 10.1177/0091217418791439. Epub 2018 Aug 4. PMID 30079814
- [Derived] Kim JM, Stewart R, Lee YS, Lee HJ, Kim MC, Kim JW, Kang HJ, Bae KY, Kim SW, Shin IS, Hong YJ, Kim JH, Ahn Y, Jeong MH, Yoon JS. Effect of Escitalopram vs Placebo Treatment for Depression on Long-term Cardiac Outcomes in Patients With Acute Coronary Syndrome: A Randomized Clinical Trial. JAMA. 2018 Jul 24;320(4):350-358. doi: 10.1001/jama.2018.9422. Erratum In: JAMA. 2018 Nov 27;320(20):2154. doi: 10.1001/jama.2018.15103. PMID 30043065
- [Derived] Kim JM, Stewart R, Kang HJ, Bae KY, Kim SW, Shin IS, Hong YJ, Ahn Y, Jeong MH, Yoon JS. BDNF methylation and depressive disorder in acute coronary syndrome: The K-DEPACS and EsDEPACS studies. Psychoneuroendocrinology. 2015 Dec;62:159-65. doi: 10.1016/j.psyneuen.2015.08.013. Epub 2015 Aug 17. PMID 26313133
- [Derived] Kim JM, Stewart R, Bae KY, Kang HJ, Kim SW, Shin IS, Hong YJ, Ahn Y, Jeong MH, Yoon JS. Correlates and Escitalopram Treatment Effects on Sleep Disturbance in Patients with Acute Coronary Syndrome: K-DEPACS and EsDEPACS. Sleep. 2015 Jul 1;38(7):1105-11. doi: 10.5665/sleep.4822. PMID 25581916
- [Derived] Kim JM, Stewart R, Bae KY, Kang HJ, Kim SW, Shin IS, Hong YJ, Ahn Y, Jeong MH, Yoon JS. Effects of depression co-morbidity and treatment on quality of life in patients with acute coronary syndrome: the Korean depression in ACS (K-DEPACS) and the escitalopram for depression in ACS (EsDEPACS) study. Psychol Med. 2015 Jun;45(8):1641-52. doi: 10.1017/S003329171400275X. Epub 2014 Nov 21. PMID 25412614
- [Derived] Kim JM, Bae KY, Stewart R, Jung BO, Kang HJ, Kim SW, Shin IS, Hong YJ, Kim JH, Shin HY, Kang G, Ahn Y, Kim JK, Jeong MH, Yoon JS. Escitalopram treatment for depressive disorder following acute coronary syndrome: a 24-week double-blind, placebo-controlled trial. J Clin Psychiatry. 2015 Jan;76(1):62-8. doi: 10.4088/JCP.14m09281. PMID 25375836